CLINICAL TRIAL: NCT03474718
Title: Evaluating the Efficacy of Platelet-rich Plasma Therapy in the Treatment of Androgenic Alopecia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00045844
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Androgenic Alopecia
Keywords: scalp; hair loss; platelet-rich plasma therapy
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Second offsite investigator will assess the patient for clinical improvement and will be unaware of the patient's randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): At the baseline visit subjects will be randomized to either group A or group B. Group A will receive PRP on left side of scalp and placebo (saline solution) on right side of scalp.
  Interventions: Biological: Platelet-rich Plasma Left Side
- Group B (Experimental): At the baseline visit subjects will be randomized to either group A or group B. Group B will receive PRP on right side of scalp and placebo (saline solution) on left side of scalp.
  Interventions: Biological: Platelet-rich Plasma Right Side

INTERVENTIONS:
Biological: Platelet-rich Plasma Left Side — Group A will receive PRP on left side of scalp and placebo (saline solution) on right side of scalp.
  Arms: Group A
Biological: Platelet-rich Plasma Right Side — Group B will receive PRP on right side of scalp and placebo (saline solution) on left side of scalp.
  Arms: Group B

SUMMARY:
The study team will assess the efficacy of platelet-rich plasma therapy, a special blood product which is from the participant's own body, in the treatment of androgenic alopecia (also known as male pattern hair loss) in females.

DETAILED DESCRIPTION:
Androgenic alopecia, or male-pattern hair loss affects both men and women. This hair loss pattern is typically characterized by thinning at the crown of scalp and/or M-shaped hair line in males or diffuse thinning throughout in females. Platelet-rich plasma (PRP) therapy has recently been studied as a hair rejuvenation therapy in patients with non-inflammatory alopecia. Though the mechanism of action is not well understood, PRP is thought to promote angiogenesis and enhance blood flow around hair follicles via platelet-derived growth factor (PDGF), transforming growth factor (TGF), and vascular endothelial growth factor (VEGF). The primary objective of the study is to determine whether PRP, administered once monthly for 3 months improves clinical outcomes and quality of life in females with androgenic alopecia. This is a randomized, placebo-controlled, double-blind, half-head, single center clinical study where sixteen subjects with androgenic alopecia will be recruited. Dermatology Life Quality Index will be assessed at several time points. Disease severity will be measured using the Severity of Alopecia Tool (SALT), Alopecia Density and Extent Score (ALODEX); Trichoscan images will be captured to document participants' clinical progress. Adverse events will be recorded at each visit, treatment will be discontinued if any subject experience a serious adverse event. Treatment visits will take place at baseline, 4 weeks (1 month), 8 weeks (2 months), and 12 weeks (3 month). A follow-up, non-treatment visit will take place at 24 weeks (6 months). The study team hypothesizes that PRP will improve DLQI, SALT, ALODEX, hair count (number of hairs/0.65 cm2), hair density (number of hairs/cm2), hair diameter, anagen to telogen ratio, and vellus hair to terminal hair ratio in female subjects with androgenic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥18 years of age at baseline visit.
* Documentation of androgenic alopecia diagnosis as evidenced by one or more clinical features
* Not currently on any treatment for alopecia, or has undergone 2-week washout period if recently on medication(s) for alopecia
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Pregnant or breastfeeding
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Have an infection, metastatic disease or certain skin conditions (ie. Psoriasis) which could worsen or spread with injections
* Diagnosed with a blood or bleeding disorder
* Diagnosed with anemia
* Currently on anticoagulant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Severity of Alopecia Tool (SALT) from baseline | 6 months
  Change in Severity of Alopecia Tool (SALT) from baseline.
  SALT scoring - This calculation is based on a scoring system. The scalp is divided into the following 4 areas:
  Vertex: 40% (0.4) of scalp surface area. Right profile of scalp: 18% (0.18) of scalp surface area. Left profile of scalp: 18% (0.18) of scalp surface area. Posterior aspect of scalp: 24% (0.24) of scalp surface area. Percentage of hair loss in any of these areas is the percentage hair loss multiplied by percent surface area of the scalp in that area.
  SALT score is the sum of percentage of hair loss in all the above-mentioned areas. For e.g., if the percentage hair loss in vertex, right profile, left profile and posterior aspect is 20, 30, 40 and 50% respecively; then, SALT score = (20 ´ 0.4) = (30 ´ 0.18) + (40 ´ 0.18) + (50 ´ 0.24) = 8+5.4+7.2+12 = 32.6 Lower score denote better outcomes.

SECONDARY OUTCOMES:
Change in Hair Count (number of hairs/0.65cm^2) | 6 months
  Change in Hair Count (number of hairs/0.65cm^2), as assessed via Trichoscan
Change in Hair Density (number of hairs/cm^2) | 6 months
  Change in Hair Density (number of hairs/cm^2), as assessed via Trichoscan

OTHER OUTCOMES:
Change in Hair Diameter | 6 months
  Change in Hair Diameter, as assessed via Trichoscan
Anagen to Telogen Ratio | 6 months
  Anagen to Telogen Ratio, as assessed via Trichoscan
Vellus Hair to Terminal Hair Ratio | 6 months
  Vellus Hair to Terminal Hair Ratio, as assessed via Trichoscan
Change in Dermatology Life Quality Index (DLQI) | 6 months
  Change in Dermatology Life Quality Index (DLQI)
  10 question are asked pertaining to symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment.
  The scoring of each answer is as follows:
  Very much scored 3 A lot scored 2 A little scored 1 Not at all scored 0 Not relevant scored 0 Question unanswered scored 0 Question 7: "prevented work or studying" scored 3 The DLQI is calculated by adding the score of each question. The maximum score is 30 and the minimum is 0. The higher the score, the more quality of life is impaired.
  Meaning of DLQI Scores 0-1 = no effect at all on patient's life 2-5 = small effect on patient's life 6-10 = moderate effect on patient's life 11-20 = very large effect on patient's life 21-30 = extremely large effect on patient's life

CONTACTS AND LOCATIONS:
Overall Officials: Rita Pichardo, MD, Principal Investigator — Wake Forest University School of Medicine, Department of Dermatology
Locations (1):
- Wake Forest University Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No